CLINICAL TRIAL: NCT03226847
Title: Pulmonary Vein Isolation in Athletes: Effects on Peak Performance and Pulmonary Vein Function
Brief Title: Pulmonary Vein Isolation in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Bryan Baranowski, Principal Investigator, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-584
Record Dates: First submitted 2017-07-20; First posted 2017-07-24 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Athletes; Atrial Fibrillation; Catheter Ablation
Keywords: Atrial Fibrillation, Athletes, Pulmonary Vein Isolation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulmonary Vein Isolation (Experimental): ablation
  Interventions: Procedure: Pulmonary Vein Isolation

INTERVENTIONS:
Procedure: Pulmonary Vein Isolation — Standard antral pulmonary vein isolation using radiofrequency ablation catheters

SUMMARY:
Pulmonary vein isolation (PVI) has become a common and effective treatment for paroxysmal and persistent atrial fibrillation (AF), particularly in patients with drug-refractory disease. Intense endurance exercise is a known risk factor for atrial fibrillation. In general, these athletes poorly tolerate most common antiarrhythmic drugs used for atrial fibrillation control and often PVI is recommended for durable management. While the efficacy of PVI in athletes is similar to the general AF population, some athletes with lone atrial fibrillation report a reduction in subjective exertional capacity following PVI, despite maintenance of sinus rhythm and absence of pulmonary vein stenosis on imaging. The investigators hypothesize that PVI may alter pulmonary vein function and affect peak exercise performance.

The investigators propose a small, prospective study of endurance athletes undergoing antral PVI for treatment of lone atrial fibrillation. Peak metabolic performance and pulmonary vein function will be assessed pre- and post-PVI by metabolic stress testing and cardiac MRI, respectively.

DETAILED DESCRIPTION:
Endurance athletes with paroxysmal or persistent atrial fibrillation undergoing primary pulmonary vein isolation will be prospectively enrolled prior to PVI.

Patients will undergo metabolic exercise stress testing as well as resting CMR 1-4 weeks prior to PVI. Metabolic stress testing and CMR will be repeated at 6 month follow-up. Quality of life questionnaires will also be collected at pre- and post-PVI visits. Metabolic treadmill stress testing will follow standard protocol and measure hemodynamics with escalating metabolic output and characterize peak exercise capacity (METs) and oxygen consumption (VO2 max).

CMR evaluation will include standard anatomic imaging of pulmonary vein and left atrial anatomy at rest. Additional cine CMR sequences willbe included for focused evaluation of dynamic pulmonary vein cross-sectional area. 3D navigator whole heart imaging and MRA (single gadolinium dose) will be obtained to measure pulmonary vein flow. CMR sequences to characterize left atrial function, including phasic volumes and emptying fractions (total, passive, active) will also be performed.

Data on heart rate variability will additionally be collected at pre- and post-PVI clinic visits, as well as the morning after PVI (hospital day 1).

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal or Persistent AF
* Endurance or highly trained athletes (>3H training/week for >10 yrs)
* NSR at time of stress testing

Exclusion Criteria:

* Structural Heart Disease; LVEF <45%
* Moderate or Severe Valvular disease
* eGFR < 30
* Contraindication to MRI
* Less than average functional capacity
* Previous episode of AF of >14 days duration
* Previous pulmonary vein isolation
* Imaging evidence of pulmonary vein stenosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
Peak Oxygen Consumption (VO2) | up to 6 months
  Assessed by cardiopulmonary stress testing

SECONDARY OUTCOMES:
Pulmonary vein function | 1-4 weeks prior to PVI. Reassessed at 6 months post-PVI.
  Change in pulmonary vein cross sectional area measured by resting cardiac MRI
Heart Rate Variability | 1-4 weeks prior to PVI. Reassessed at 1 day and 6 months post-PVI.
  Time and frequency domain analysis of subjects heart rate variability using 5- minute protocol
Subjective Assessment of Athletic Performance | 1-4 weeks prior to PVI. Reassessed at 6 months post-PVI.
  Measured by athlete-specific questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Baranowski, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calvo N, Mont L, Tamborero D, Berruezo A, Viola G, Guasch E, Nadal M, Andreu D, Vidal B, Sitges M, Brugada J. Efficacy of circumferential pulmonary vein ablation of atrial fibrillation in endurance athletes. Europace. 2010 Jan;12(1):30-6. doi: 10.1093/europace/eup320. PMID 19923171